CLINICAL TRIAL: NCT04011033
Title: Study of Adoptive Transfer of Invariant Natural Killer T Cells Combined With TAE/TACE to Treat Unresectable Hepatocellular Carcinoma (HCC): Phase II Clinical Trial
Brief Title: Study of Adoptive Transfer of iNKT Cells Combined With TAE/TACE to Treat Unresectable HCC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing YouAn Hospital (Other)
Collaborators: Beijing Shijitan Hospital, Capital Medical University (Other); Beijing Ditan Hospital (Other)
Responsible Party: Principal Investigator, LU JUN, Director of Hepatology and Cancer Biotherapy Ward, Beijing YouAn Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Beijing Youan Ethics [2018]016
Record Dates: First submitted 2019-07-03; First posted 2019-07-08 (Actual); Results first posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-09

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Interleukin-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAE/TACE+iNKT for unresectable HCC (Experimental): TAE/TACE combined with autologous iNKT cells infusion will be applied for patients in experimental group. TAE/TACE will be performed at 0th and 4th week. 5×10^8-10^9/m2 iNKT cells will be infused to patients at 1st, 3rd, 5th, 7th, 9th, 11th week after first TAE/TACE therapy.
  Interventions: Biological: iNKT cells; Drug: Human recombinated Interleukin-2; Procedure: TAE/TACE
- TAE/TACE for unresectable HCC (Other): TAE/TACE will be conducted at 0th week and 4th week.
  Interventions: Procedure: TAE/TACE

INTERVENTIONS:
Biological: iNKT cells — 5×10^8-10^9/m2 iNKT cells will be infused to patients at 1st, 3rd, 5th, 7th, 9th, 11th week after first TAE/TACE therapy.
  Other Names: invariant Natural Killer T cells
  Arms: TAE/TACE+iNKT for unresectable HCC
Drug: Human recombinated Interleukin-2 — IL-2 will be given at a dose of 25,000 IU/kg/day for 5-14 days after iNKT cells infusion.
  Other Names: IL-2
  Arms: TAE/TACE+iNKT for unresectable HCC
Procedure: TAE/TACE — TAE/TACE will be conducted to all patients at 0th week and 4th week.
  Other Names: Transcatheter Arterial embolization/Transcatheter Arterial chemoembolization

SUMMARY:
Hepatocellular carcinoma (HCC) is a common disease with high mortality. More than 80% patients receive a diagnosis when their tumors are too advanced for curative approaches and have a dismal prognosis. invariant Natural Killer T (iNKT) cell exhibit antitumor activity against malignant tumors through producing high levels of cytokines. iNKT cells are abundant in the liver, but their function is defective in liver cancer. After expansion and restored function in vitro, iNKT cells can home to liver, then they play key antitumor function. We have finished a phase I study of adoptive transfer of autologous iNKT cells for treating patients with unresectable HCC. Safety and feasibility of iNKT infusion was proved. The purpose of this study was to verify the effectiveness of iNKT cell infusion in patients with unresectable HCC who had previously failed transcatheter arterial embolization (TAE) / transcatheter arterial chemoembolization (TACE).

DETAILED DESCRIPTION:
Patients with unresectable HCC will be enrolled and divided into two groups. Patients in trial group will be treated with combination of TAE/TACE and adoptive transfer of autologus iNKT cells. TAE/TACE will be performed at 0th and 4th week. iNKT cells will be infused at 1st, 3rd, 5th, 7th, 9th, 11th week after first TAE/TACE therapy. Patients in control group will be treated with TAE/TACE at 0th and 4th week. Overall survival (OS) time, progression-free survival (PFS) time, objective response rate(ORR), disease control rate(DCR) will be monitored.

According to JSH guidelines, TAE/TACE failure is defined as an insufficient response after ≧2 consecutive TAE/TACE procedures that is evident on response evaluation computed tomography or magnetic resonance imaging after 1-3 months, these patients do not respond sufficiently to TAE/TACE.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years.
* Patients with hepatocellular carcinoma (BCLC, stageB/C) proved by histopathology or proved by CT or MRI imaging system, relapsed after previous therapy and no effective therapies known at this time.
* Life expectancy of ≥ 12 weeks.
* WBC>3.0×10^9/L, LYMPH> 0.8×10^9/L, Hb>85g/L, PLT>50×10^9/L, Cre<1.5×the upper limit of normal value.
* iNKT>10 cell/mL in peripheral blood mononuclear cell (PBMC).
* Able to understand and sign the informed consent.

Exclusion Criteria:

* Any uncontrolled systematic disease: hypertension, heart disease, and et al.;
* Portal vein tumor thrombus, central nervous system tumor metastasis, or combined with other tumors;
* Receiving radiochemotherapy, local therapy, or targeting drugs within 4 weeks prior to this treatment;
* Unstable immune systematic diseases or infectious diseases;
* Combined with AIDS or syphilis;
* Patients with history of stem cell or organ transplantation;
* Patients with allergic history to related drugs and immunotherapy;
* Patients with complications associated with liver diseases: moderate or severe pleural effusion, pericardial effusion, ascites, or gastrointestinal hemorrhage;
* Pregnant or lactating subjects;
* Unsuitable subjects considered by clinicians.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2023-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jun Lu, Director, Study Chair — Beijing YouAn Hospital
Locations (1):
- Beijing Youan Hospital,Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Guo J, Bao X, Liu F, Guo J, Wu Y, Xiong F, Lu J. Efficacy of Invariant Natural Killer T Cell Infusion Plus Transarterial Embolization vs Transarterial Embolization Alone for Hepatocellular Carcinoma Patients: A Phase 2 Randomized Clinical Trial. J Hepatocell Carcinoma. 2023 Aug 21;10:1379-1388. doi: 10.2147/JHC.S416933. eCollection 2023. PMID 37637501

RESULTS

PARTICIPANT FLOW:
Groups:
- TAE/TACE+iNKT for Unresectable HCC: TAE/TACE combined with autologous iNKT cells infusion will be applied for patients in experimental group. TAE/TACE will be performed at 0th and 4th week. 5×10^8-10^9/m2 iNKT cells will be infused to patients at 1st, 3rd, 5th, 7th, 9th, 11th week after first TAE/TACE therapy.
  iNKT cells: 5×10^8-10^9/m2 iNKT cells will be infused to patients at1st, 3rd, 5th, 7th, 9th, 11th week after first TAE/TACE therapy.
  Human recombinated Interleukin-2: IL-2 will be given at a dose of 25,000 IU/kg/day for 5-14 days after iNKT cells infusion.
  TAE/TACE: TAE/TACE will be conducted to all patients at 0th week and 4th week.
Period: Overall Study
Arm/Group | TAE/TACE+iNKT for Unresectable HCC | TAE/TACE for Unresectable HCC
Started | 30 | 30
Completed | 27 | 27
Not Completed | 3 | 3
Not completed — Physician Decision | 2 | 3
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- TAE/TACE+iNKT for Unresectable HCC: TAE/TACE combined with autologous iNKT cells infusion will be applied for patients in experimental group. TAE/TACE will be performed at 0th and 4th week. 5×10^8-10^9/m2 iNKT cells will be infused to patients 1st, 3rd, 5th, 7th, 9th, 11th week after first TAE/TACE therapy.
  iNKT cells: 5×10^8-10^9/m2 iNKT cells will be infused to patients at 1st, 3rd, 5th, 7th, 9th, 11th week after first TAE/TACE therapy.
  Human recombinated Interleukin-2: IL-2 will be given at a dose of 25,000 IU/kg/day for 5-14 days after iNKT cells infusion.
  TAE/TACE: TAE/TACE will be conducted to all patients at 0th week and 4th week.
- Total: Total of all reporting groups
Arm/Group | TAE/TACE+iNKT for Unresectable HCC | TAE/TACE for Unresectable HCC | Total
Number analyzed (Participants) | 27 | 27 | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 21 | 40
  >=65 years | 8 | 6 | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 23 | 24 | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 27 | 27 | 54
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 27 | 27 | 54
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  China | 27 | 27 | 54

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival(PFS)
Description: PFS is the duration from the date of enrolled into clinical trial to the date of first documentation of tumor progression.
  Progression is defined using Modified RECIST (mRECIST),as an increase of at least 20% in the sum of the diameters of viable (enhancing) target lesions, taking as reference the smallest sum of the diameters of viable (enhancing) target lesions recorded since treatment started.
Time Frame: From date of enrollment to disease progression according to mRECIST, or death from any cause, whichever occurred first，approximately 2 years.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- TAE/TACE+iNKT for Unresectable HCC: TAE/TACE combined with autologous iNKT cells infusion will be applied for patients in experimental group. TAE/TACE will be performed at 0th and 4th week. 5×10^8-10^9/m2 iNKT cells will be infused to patients at 1st, 3rd, 5th, 7th, 9th, 11th week after first TAE/TACE therapy.
  iNKT cells: 5×10^8-10^9/m2 iNKT cells will be infused to patients at 1st, 3rd, 5th, 7th, 9th, 11th week after first TAE/TACE therapy. therapy.
  Human recombinated Interleukin-2: IL-2 will be given at a dose of 25,000 IU/kg/day for 5-14 days after iNKT cells infusion.
  TAE/TACE: TAE/TACE will be conducted to all patients at 0th week and 4th week.
Arm/Group | TAE/TACE+iNKT for Unresectable HCC | TAE/TACE for Unresectable HCC
Number analyzed (Participants) | 27 | 27
months | 5.7 [4.3 to 7.0] | 2.7 [2.3 to 3.2]
Statistical Analysis 1: Comparison: TAE/TACE+iNKT for Unresectable HCC vs TAE/TACE for Unresectable HCC; Test type: Other; p < 0.001, Log Rank; Hazard Ratio (HR) = 0.32, 95% CI 2-sided [0.16 to 0.63]

2. Secondary Outcome: Overall Survival(OS)
Description: OS is the duration from the date of enrollment to the date of death due to any causes.
Time Frame: From date of randomization until the date of death from any cause, whichever came first, assessed up to 60 months.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | TAE/TACE+iNKT for Unresectable HCC | TAE/TACE for Unresectable HCC
Number analyzed (Participants) | 27 | 27
months | 25.9 [12.4 to 44.4] | 17.3 [7.5 to 27.6]

3. Secondary Outcome: Objective Response Rate(ORR)
Description: ORR is the proportion of patients who had a response rate including complete remission (CR) and partial remission (PR) evaluated by imaging according to mRECIST for target lesions and assessed by MRI/CT: Complete Response (CR), Disappearance of any intratumoral arterial enhancement in all target lesions；Partial Response (PR), At least a 30% decrease in the sum of diameters of viable (enhancement in the arterial phase) target lesions, taking as reference the baseline sum of the diameters of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Evaluation was performed at the 12th week after the start of the treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | TAE/TACE+iNKT for Unresectable HCC | TAE/TACE for Unresectable HCC
Number analyzed (Participants) | 27 | 27
Participants | 14 | 3
Statistical Analysis 1: Comparison: TAE/TACE+iNKT for Unresectable HCC vs TAE/TACE for Unresectable HCC; Test type: Other; p = 0.003, Fisher Exact

4. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR is the proportion of patients who had a response rate including complete remission (CR), partial remission (PR) and disease stabilization (SD) evaluated by imaging according to mRECIST for target lesions and assessed by MRI/CT: Complete Response (CR), Disappearance of any intratumoral arterial enhancement in all target lesions；Partial Response (PR), At least a 30% decrease in the sum of diameters of viable (enhancement in the arterial phase) target lesions, taking as reference the baseline sum of the diameters of target lesions;Stable disease(SD), Any cases that do not qualify for either partial response or progressive disease. Disease Control Rate (DCR) = CR + PR + SD.
Time Frame: Evaluation was performed at the 12th week after the start of the treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | TAE/TACE+iNKT for Unresectable HCC | TAE/TACE for Unresectable HCC
Number analyzed (Participants) | 27 | 27
Participants | 23 | 9
Statistical Analysis 1: Comparison: TAE/TACE+iNKT for Unresectable HCC vs TAE/TACE for Unresectable HCC; Test type: Other; p < 0.001, Fisher Exact

5. Secondary Outcome: Adverse Events(AEs)
Description: The severities of AEs will be divided into 5 levels according to the National Cancer Institute (NCI) Common Terminology Standard for Adverse Events (CTCAE) version 4.03.
Time Frame: The occurrence of AEs was observed for an average of 24 weeks after the completion of treatment (between 0-11 weeks of treatment) for up to a 60 week period in total.
Measure: Count of Participants; unit: Participants
Arm/Group | TAE/TACE+iNKT for Unresectable HCC | TAE/TACE for Unresectable HCC
Number analyzed (Participants) | 27 | 27
Participants
  Chill (Any Grade) | 0 | 0
  Chill (≧ Grade 3) | 0 | 0
  Fatigue(Any Grade) | 3 | 5
  Fatigue(≧ Grade 3) | 0 | 0
  Fever (Any Grade) | 3 | 5
  Fever (≧ Grade 3) | 0 | 0
  Injection site reaction(Any Grade) | 0 | 0
  Injection site reaction (≧ Grade 3) | 0 | 0
  Callosity(Any Grade) | 4 | 0
  Callosity(≧ Grade 3) | 0 | 0
  Activation time of partial prothrombin (Any Grade) | 0 | 0
  Activation time of partial prothrombin (≧ Grade 3) | 0 | 0
  Alanine aminotransferase increased (Any Grade) | 1 | 8
  Alanine aminotransferase increased (≧ Grade 3) | 0 | 2
  Aspartate aminotransferase increased (Any Grade) | 4 | 5
  Aspartate aminotransferase increased (≧ Grade 3) | 0 | 0
  Blood bilirubin increased (Any Grade) | 3 | 6
  Blood bilirubin increased (≧ Grade 3) | 0 | 2
  Alkaline phosphatase increased (Any Grade) | 1 | 2
  Alkaline phosphatase increased (≧ Grade 3) | 0 | 0
  Glutamyl transpeptidase increased (Any Grade) | 6 | 6
  Glutamyl transpeptidase increased (≧ Grade 3) | 1 | 1
  Cholesterol high(Any Grade) | 1 | 1
  Cholesterol high(≧ Grade 3) | 0 | 0

6. Secondary Outcome: Time to Quality of Life (QoL) Deterioration
Description: EORTC QLQ-C30: European Organization for Research on Treatment of Cancer Quality of Life Questionnare-Core 30.
  The totally 30 items spread out over five functional scales (15 items), three symptom scales (7 items), a global health status/QoL scale (2 items), and six single items. 1-28 item ranges 1: not at all, 2: a little, 3: quite a lit, 4: very much; 29-30 item ranges 1-7 from very poor to excellent. Raw score (RS) is an average of all items in each area. Standardized score is in the range of 0-100 by formula SS=[1-(RS-1)/n] x100 (function) or SS=[（RS-1）/n]x100 (symptom or overall health) respectively. A high scale score represents a higher/healthy response level.
  Time to deterioration was defined as a decrease from baseline of 10 points or more on the EORTC QLQ-C30 maintained for two consecutive assessments.
Time Frame: Data will be collected at baseline and every 4 weeks until disease progression, then every 8 weeks for up to 60 weeks.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | TAE/TACE+iNKT for Unresectable HCC | TAE/TACE for Unresectable HCC
Number analyzed (Participants) | 27 | 27
months | 9.2 [6.0 to 13.3] | 3.0 [2.9 to 3.0]
Statistical Analysis 1: Comparison: TAE/TACE+iNKT for Unresectable HCC vs TAE/TACE for Unresectable HCC; Test type: Other; p = 0.001, Log Rank; Hazard Ratio (HR) = 0.37, 95% CI 2-sided [0.19 to 0.71]

ADVERSE EVENTS:
Time Frame: The occurrence of AEs was observed for an average of 24 weeks after the completion of treatment (between 0-11 weeks of treatment) for up to a 60 week period in total.
Arm/Group | TAE/TACE+iNKT for Unresectable HCC | TAE/TACE for Unresectable HCC
All-Cause Mortality (participants affected / at risk) | 5/27 | 4/27
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/27
Other Adverse Events (participants affected / at risk) | 14/27 | 15/27
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TAE/TACE+iNKT for Unresectable HCC (N=27) | TAE/TACE for Unresectable HCC (N=27)
Fatigue (General disorders) | 3 (3) | 5 (5)
Fever (General disorders) | 3 (3) | 5 (5)
Callosity (General disorders) | 4 (4) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 8 (8)
Aspartate aminotransferase increased (Investigations) | 4 (4) | 5 (5)
Blood bilirubin increased (Investigations) | 3 (3) | 6 (6)
Alkaline phosphatase increased (Investigations) | 1 (1) | 2 (2)
Glutamyl transpeptidase increased (Investigations) | 6 (6) | 6 (6)
Cholesterol high (Investigations) | 1 (1) | 1 (1)

LIMITATIONS AND CAVEATS:
One limitation of our study is that patients only received two cycles of TAE and the duration of iNKT therapy was only 3 months; thus, our study was not long enough to adequately assess OS. A second limitation was the small sample size, but our promising data prompts future studies in larger cohorts to more thoroughly delineate how iNKT cell therapy can be used in the context of TACE/TAE to improve therapeutic options for patients with unresectable HCC.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-01): https://cdn.clinicaltrials.gov/large-docs/33/NCT04011033/Prot_SAP_000.pdf